CLINICAL TRIAL: NCT05035706
Title: Anti-Leukemia Immune Responses After Irradiation of Extramedullary Tumors
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0037; NCI-2021-08685 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0037 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-25; First posted 2021-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia; Myeloid Leukemia; Recurrent Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myeloid | interventions — Biopsy; Photography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (biopsy, biospecimen collection) (Experimental): Patients undergo biopsy prior to radiation therapy and 7-14 days after radiation therapy. Patients also undergo blood sample collection prior to therapy (within 7 days of starting radiation therapy), 1 and 7 days post completion of radiation therapy. Patients' photographs of the biopsy site are taken before and at 4-6 weeks post completion of radiation, and their medical records are reviewed for up to 2 years.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Photography

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood and tissue sample collection
  Other Names: Biological Sample Collection
Other: Electronic Health Record Review — Medical records reviewed
Other: Photography — Photographs taken

SUMMARY:
This clinical trial assesses how the immune system responds to leukemia tumors after low dose radiation delivered as part of standard of care. The information learned in this study may help them know if adding immunotherapy (a type of treatment that uses the immune system to fight cancer) can be helpful in future leukemia patients receiving radiation.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify changes in anti-leukemia immune responses after local radiotherapy to extramedullary sites.

II. Develop an annotated biospecimen panel of extramedullary leukemia biopsies prior to and after radiotherapy to examine local immune responses using transcriptional profiling, immunofluorescence and single cell analyses.

III. Define changes in the T cell receptor (TCR) clonotypes, functionality and inflammatory cytokine levels in peripheral blood leukocytes and serum.

IV. Correlate changes in anti-tumor immune responses with clinic-pathological variables and patient outcomes.

SECONDARY OBJECTIVES:

I. To assess the overall response rate (ORR= complete response [CR] + partial response [PR]) of the extramedullary tumor treated with radiation therapy.

II. To assess the CR of extramedullary tumor treated with radiation therapy. III. Determine the duration of response (DOR), event-free survival (EFS).

OUTLINE:

Patients undergo biopsy prior to radiation therapy and 7-14 days after radiation therapy. Patients also undergo blood sample collection prior to therapy (within 7 days of starting radiation therapy), 1 and 7 days post completion of radiation therapy. Patients' photographs of the biopsy site are taken before and at 4-6 weeks post completion of radiation, and their medical records are reviewed for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with new or recurrent myeloid leukemia
* Aged >= 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status < 4
* Patient have measurable and amenable to biopsy under local anesthesia without the need for imaging directed procedure
* Ability to understand and provide signed informed consent
* Females must be surgically or biologically sterile or postmenopausal (amenorrhoeic for at least 12 months) or if of childbearing potential, must have a negative serum or urine pregnancy test within 72 hours before the start of the treatment. Women of childbearing potential must agree to use an adequate method of contraception during the study and until the last radiation treatment. Males must be surgically or biologically sterile or agree to use an adequate method of contraception during the study and until the last radiation treatment

Exclusion Criteria:

* Patients who are unwilling to participate
* Patients unwilling to undergo the biopsy before or after radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Changes in anti-leukemia immune responses | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bouthaina S Dabaja, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org